CLINICAL TRIAL: NCT05680194
Title: Prospective Research for Elderly (≥65 Years Old) Early Breast Cancer Patients
Acronym: EEBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EEBC
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female
Keywords: ≥65 Years Old; early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy; Radiotherapy; Diphosphonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paraffin section
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: operation — operation methods: breast-conserving surgery, mastectomy, axillary lymph node dissection, sentinal lymphnodes biopsy; chemotherapy regimens: AC, TC, AC-T/P, TCrb, TAC, capecitabine; ovarian protection:GnRHa; endocrine therapy: Aromatase inhibitor, TAM, Fulvestrant, CDK4/6 inhibitors; target therapy: trastuzumab，patuzumab, Pyrotinib.
  Other Names: chemotherapy; radiotherapy; endocrine therapy; targeted therapy
Drug: Bisphosphonate — Bisphosphonate

SUMMARY:
The elderly patients over 65 years old with breast cancer have concomitant diseases, poor tolerance to conventional treatment, and the specific prognosis of breast cancer is relatively good. Previous studies on breast cancer have almost excluded elderly breast cancer patients, and conventional treatment schemes cannot meet the clinical diagnosis and treatment needs of elderly breast cancer patients. The establishment of a prognosis model for elderly breast cancer patients can provide personalized treatment programs. This is important for prolonging the survival time of patients and improving the quality of life. This project plans to observe the relationship between prognosis and pathological staging, molecular typing, and concomitant diseases of elderly breast cancer patients in combination with immune genes, and establish a prognosis model of elderly breast cancer and verify it. This project is expected to establish a new prognostic model for elderly breast cancer patients, accurately judge the prognosis of patients, and provide a new basis for hierarchical and personalized treatment of elderly breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* female patients with breast cancer
* ≥65 Years Old
* patients with breast cancer received operation in Peking Union Medical College Hospital
* treatment regimen was made in Peking Union Medical College Hospital

Exclusion Criteria:

* patients with metastasis
* patietns with recurrence
* patients without pathological information

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: the patients ≥65 Years Old with breast cancer who received operaion in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
5-y DFS | 5 year
  5-years of disease free survival
5-y BCSS | 5 year
  5-year of breast cancer-specific survival

SECONDARY OUTCOMES:
5-y OS | 5 year
  5-year overall survival
10-y DFS | 10 year
  10-years of disease free survival
10-y BCSS | 10 year
  10-year of breast cancer-specific survival
10-y OS | 10 year
  10-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No